CLINICAL TRIAL: NCT03646942
Title: Evaluation of Low-Level-LASER Therapy (LLLT) Effect on Accelerating Orthodontic Tooth Movement For Crowded Upper Incisors Leveling and Alignment in Lingual Orthodontic Patients: A Randomized Clinical Controlled Trial
Brief Title: The Role of Low Level Laser Therapy in Acceleration of Teeth Alignment in Lingual Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-08-2018
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion, Angle Class I; Crowding
MeSH Terms: conditions — Malocclusion, Angle Class I; Crowding | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lingual orthodontics (Active Comparator): Patients will be treated with lingual braces without being irradiation with low level laser therapy. Treatment will go forward in the normal manner. Archwires will be changed in the traditional way.
  Interventions: Radiation: low level laser therapy; Device: Lingual Orthodontics
- Low level laser therapy (Experimental): Patients will be subjected to low level laser therapy during their orthodontic treatment using lingual braces.
  Interventions: Radiation: low level laser therapy

INTERVENTIONS:
Radiation: low level laser therapy — low level laser therapy will be used in order to induce tooth movement. low level laser with a wave length of 830 nm, output of 150 mw, energy of 2 j per point and application time of 15 seconds per point will be applied on each tooth of the six upper incisors according to this protocol: the root will be divided into 2 halves; gingival and cervical. Laser will be applied in the center of each half from both the buccal and palatal sides which means 4 application points and a total energy of 8 Joules/each tooth.
  Other Names: LLLT; soft tissue laser
Device: Lingual Orthodontics — Lingual braces will be used to conduct the orthodontic treatment of patients with moderate level of crowding on the upper dental arch.
  Arms: Lingual orthodontics

SUMMARY:
We will treat patients with class I malocclusion who have moderate crowding (4-6 mm) according to Little's irregularity index and asses the efficacy of low level laser therapy in accelerating orthodontic tooth movement .

There is two groups :

1. treated with Low level laser therapy (LLLT)
2. treated traditionally without any irradiation Patients will be randomly allocated in any group and all data will be collected through photographs when leveling and alignment completed.

Also pain levels will be assessed using numeric rating scale to compare between the two groups and if laser really can relief pain or not .

DETAILED DESCRIPTION:
The time of orthodontic treatment is considered to be one of the most concerns for patients. The study will investigate the effect of low level laser therapy on the speed of orthodontic tooth movement during the correction of moderately crowded anterior upper teeth using lingual orthodontic appliance.

The study will be accomplished with two arms, the first is LLLT arm and the other is the control arm without any active intervention.

Low level laser with a wave length of 830 nm, output of 150 mW, energy of 2 J per point and application time of 15 seconds per point will be applied on each tooth of the six upper incisors according to this protocol: the root will be divided into 2 halves; gingival and cervical. Laser will be applied in the center of each half from both the buccal and palatal sides which means 4 application points and a total energy of 8 j per each tooth.

Within the limits of our knowledge, this is the first study in the world that will study acceleration of orthodontic tooth movement with lingual orthodontic .

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with mild to moderate crowding
* Old between 17-27 years
* Good oral hygiene
* Patients should be fit and well
* 4-6 mm crowding in upper incisors according to Little's index
* Enough clinical crowns length

Exclusion Criteria:

* Patients who had an old orthodontic treatment
* People who have any drug or disease affect orthodontic movement
* Any contraindication for orthodontic treatment

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Duration of tooth alignment | When the treatment is completed (i.e. tooth alignment is achieved) and this is expected to take 100 days on average
  Days required to complete tooth alignment will be counted.
Change in Tooth Alignment at one month | T1: one day before the beginning of treatment; T2: at 30 days after the onset of treatment.
  Little's Index of Irregularity will be measured at 30 days after the onset of treatment.
  This index is measured on intraoral photographs of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.
Change in Tooth Alignment at two months | T1: one day before the beginning of treatment; T2: at 60 days after the onset of treatment.
  Little's Index of Irregularity will be measured at 60 days after the onset of treatment.
  This index is measured on intraoral photographs of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.
Change in Tooth Alignment at the end of Alignment Stage | T1: one day before the beginning of treatment; T2: when alignment of teeth is complete and this is expected to occur within 90 - 120 days
  Little's Index of Irregularity will be measured when a complete alignment is achieved; this is expected between 90 to 120 days after the onset of treatment.
  This index is measured on intraoral photographs of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.

SECONDARY OUTCOMES:
Change in the levels of pain and discomfort | T1: 10 minutes following the insertion of the first wire in the beginning of treatment; T2: at 24 hours post-commencement; T3: at 48 hours; T4: at 72 hours following the placement of primary archwire
  Assessment will be performed using questionnaires via numeric rating scales (NRS) These levels will be assessed during the first stage of leveling and alignment.
Change in Patients' Acceptance | (1) one day following the beginning of the treatment, (2) after one week of the beginning of treatment, (3) after 4 weeks, (5) at the end the alignment stage which is expected to occur within 3 to 4 months
  Assessment will be performed using a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, SYRIA; Wael Al-Rasheed Omer, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus Dental School, Damascus, SYRIA; Wael Mahdi, DDS MSc PhD, Study Director — Associate Professor of Periodontics, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Orthodontic Department, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlSayed Hasan MMA, Sultan K, Hamadah O. Low-level laser therapy effectiveness in accelerating orthodontic tooth movement: A randomized controlled clinical trial. Angle Orthod. 2017 Jul;87(4):499-504. doi: 10.2319/062716-503.1. Epub 2016 Nov 21. PMID 27869476
- [Background] Khattab TZ, Farah H, Al-Sabbagh R, Hajeer MY, Haj-Hamed Y. Speech performance and oral impairments with lingual and labial orthodontic appliances in the first stage of fixed treatment. Angle Orthod. 2013 May;83(3):519-26. doi: 10.2319/073112-619.1. Epub 2012 Oct 18. PMID 23075062
- [Background] Fritz U, Diedrich P, Wiechmann D. Lingual technique--patients' characteristics, motivation and acceptance. Interpretation of a retrospective survey. J Orofac Orthop. 2002 May;63(3):227-33. doi: 10.1007/s00056-002-0124-3. English, German. PMID 12132310
- [Background] Gkantidis N, Mistakidis I, Kouskoura T, Pandis N. Effectiveness of non-conventional methods for accelerated orthodontic tooth movement: a systematic review and meta-analysis. J Dent. 2014 Oct;42(10):1300-19. doi: 10.1016/j.jdent.2014.07.013. Epub 2014 Jul 27. PMID 25072362
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Camacho AD, Velasquez Cujar SA. Dental movement acceleration: Literature review by an alternative scientific evidence method. World J Methodol. 2014 Sep 26;4(3):151-62. doi: 10.5662/wjm.v4.i3.151. eCollection 2014 Sep 26. PMID 25332914